CLINICAL TRIAL: NCT00167206
Title: A Study of Thymic Shielding in Recipients of Total Body Irradiation, Cyclophosphamide, and Fludarabine Followed by Alternate Donor Hematopoietic Stem Cell Transplantation in Patients With Fanconi Anemia
Brief Title: Stem Cell Transplantation for Fanconi Anemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Treatment with thymic shielding found safe, another study started.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0312M54991; MT2003-18 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Fanconi Anemia
Keywords: Stem Cell Transplant; Thymic Shielding; Total Body Irradiation; Chemotherapy
MeSH Terms: conditions — Fanconi Anemia | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Whole-Body Irradiation; Radiotherapy; CF regimen; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HSCT Patients (Experimental): Patients who received total body irradiation (450 cGy [centigray]) with thymic shielding prior to chemotherapy regimen and Hematopoietic Stem Cell Transplant (HSCT)
  Interventions: Procedure: Hematopoietic Stem Cell Transplant; Procedure: Thymic Shielding During Radiation; Procedure: Total Body Irradiation; Drug: Cyclophosphamide, Fludarabine

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Transplant — Bone marrow failure may be treated by giving patients stem cells that come from someone else. This is called a stem-cell transplant. As part of the transplant process, patients receive high doses of chemotherapy and/or radiation to treat their underlying disease. As one of its effects, this treatment also kills the healthy stem cells that are already in the marrow. The transplant provides new stem cells for the patient from a healthy donor; that replace the bone marrow and allow the blood counts to recover.
  Other Names: Bone Marrow Transplant
Procedure: Thymic Shielding During Radiation — protecting the thymus during total body radiation (450 cGy administered)
  Other Names: TBI
Procedure: Total Body Irradiation — Six days before the stem cells are given (day -6), subjects will receive total body irradiation with thymic shielding. Thymic shielding is done by placing a piece of lead on the chest during the irradiation treatment so that the irradiation beams do not go to the thymus.
  Other Names: Radiation Therapy, Therapuetic Radiation
Drug: Cyclophosphamide, Fludarabine — Day -5 through Day -2, subjects will receive a chemotherapy regimen of Fludarabine, Cyclophosphamide via central line
  Other Names: Cytoxan, Fludara

SUMMARY:
The purpose of this study is to determine whether thymic shielding during total body irradiation can be given and whether it will reduce the risk of infections in Fanconi Anemia patients undergoing alternate donor (not a matched sibling) stem cell transplants.

DETAILED DESCRIPTION:
All subjects will be given the same treatment regimen of total body irradiation (TBI), Fludarabine, Cyclophosphamide, and anti-thymocyte globulin (ATG), followed by an alternate donor stem cell transplant. Since this treatment regimen has been given before, without thymic shielding, we will compare the outcomes of these patients with the historical data from subjects who did not receive thymic shielding.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be less than (<) 18 years of age with a diagnosis of Fanconi anemia.
* Patients must have an HLA-A, B, DRB1 identical unrelated donor or less than or equal to (≤)1 antigen mismatched related (non-HLA-matched sibling) or <1 antigen mismatched unrelated UCB donor. Patients and donors will be typed for HLA-A and B using serological or molecular techniques and for DRB1 using high resolution molecular typing.
* Patients with FA must have aplastic anemia (AA), myelodysplastic syndrome without excess blasts, or high risk genotype as defined below.

  * Aplastic anemia is defined as having at least one of the following when not receiving growth factors or transfusions
  * Platelet count <20 x 10^9/L
  * ANC <5 x 10^8/L
  * Hgb <8 g/dL
  * Myelodysplastic syndrome with multilineage dysplasia with or without chromosomal anomalies
  * High risk genotype (e.g. IVS-4 or exon 14 FANCC mutations, or BRCA1 or 2 mutations)
* Adequate major organ function including

  * Cardiac: ejection fraction greater than (>)45%
  * Hepatic: bilirubin, AST/ALT, ALP <2 x normal
  * Karnofsky performance status >70% or Lansky performance status >50%
* Women of child-bearing age must be using adequate birth control and have a negative pregnancy test

Exclusion Criteria:

* Available HLA-genotypically identical related donor
* History of gram negative sepsis or systemic fungal infection (proven or suspected based on radiographic studies)
* Refractory anemia with excess blasts, or leukemia
* Active central nervous system (CNS) leukemia at time of hematopoietic cell transplant (HCT)
* History of squamous cell carcinoma of the head/neck/cervix within 2 years of HCT
* Pregnant or lactating female
* Prior radiation therapy preventing use of total body irradiation (TBI) 450 centigray (cGy)

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2004-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret MacMillan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] MacMillan ML, DeFor TE, Young JA, Dusenbery KE, Blazar BR, Slungaard A, Zierhut H, Weisdorf DJ, Wagner JE. Alternative donor hematopoietic cell transplantation for Fanconi anemia. Blood. 2015 Jun 11;125(24):3798-804. doi: 10.1182/blood-2015-02-626002. Epub 2015 Mar 30. PMID 25824692

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent-To-Treat: All patients with Fanconi anemia who received thymic shielding during total body irradiation (450 cGy).
Period: Overall Study
Arm/Group | Intent-To-Treat
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Exhibited Hematopoietic Recovery and Engraftment
Description: Calculated from Day 1 of hematopoietic cell transplant to Day 42 post-transplant. Hematopoietic recovery and engraftment is defined as the first of three consecutive days the patient's absolute neutrophil count is greater than or equal to 0.5X10^9/Liter.
Time Frame: Day 42 after hematopoietic cell transplant
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Participants | 15

2. Secondary Outcome: Number of Patients Who Exhibited Secondary Graft Failure
Description: Calculated from Day 1 of hematopoietic cell transplant to Day 100 after transplant. A complication after Bone Marrow Transplant in which the transplanted stem cells do not grow in the recipient's bone marrow and thus do not produce new blood cells.
Time Frame: Day 100 after hematopoietic cell transplant
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Participants | 1

3. Secondary Outcome: Number of Patients With Acute Graft Versus-Host Disease (aGVHD)
Description: Calculated from Day 1 of hematopoietic cell transplant to Day 100 after transplant. GVHD is a common complication of allogeneic bone marrow transplantation in which functional immune cells in the transplanted marrow recognize the recipient as "foreign" and mount an immunologic attack.
Time Frame: Day 100 after hematopoietic cell transplant
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Participants | 8

4. Secondary Outcome: Number of Patients With Chronic Graft Versus-Host Disease (GVHD)
Description: Calculated from Day 1 of hematopoietic cell transplant to 1 year after transplant. GVHD is a common complication of allogeneic bone marrow transplantation in which functional immune cells in the transplanted marrow recognize the recipient as "foreign" and mount an immunologic attack.
Time Frame: 1 year after hematopoietic cell transplant
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Participants | 2

5. Secondary Outcome: Number of Patients Who Exhibited Regimen-related Toxicity (RRT)
Description: Calculated from Day 1 of hematopoietic cell transplant to 1 year after transplant. Regimen-related toxicity involves harmful effects in an organism through exposure to the treatment given.
Time Frame: 1 year after hematopoietic cell transplant
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Participants | 5

6. Secondary Outcome: Immune Reconstitution - Mean Value (1 Year)
Description: Calculated mean value of patient CD4 values collected at intervals from Day 30 through 1 year post-transplant.
Time Frame: 1 year post-transplant.
Measure: Mean (Standard Deviation); unit: Number of CD4 cells per microliter
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Number of CD4 cells per microliter | 860 (870)

7. Secondary Outcome: Immune Reconstitution - Mean Value (2 Years)
Description: Calculated mean value of patient CD4 values collected at intervals from Day 30 through 2 years post-transplant.
Time Frame: at 2 years after transplant
Measure: Mean (Standard Deviation); unit: Number of CD4 cells per microliter
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Number of CD4 cells per microliter | 1100 (510)

8. Secondary Outcome: Number of Patients Alive at 1 Year
Description: Calculated from Day 1 of hematopoietic cell transplant to 1 year post-transplant.
Time Frame: 1 year after transplant
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Participants | 11

9. Secondary Outcome: Number of Patients Alive at 2 Years
Description: Calculated from Day 1 of hematopoietic cell transplant to 2 years post-transplant.
Time Frame: 2 years after transplant
Measure: Number; unit: Participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 16
Participants | 10

ADVERSE EVENTS:
Time Frame: Start of study through 1 year after transplant.
Description: Adverse events were not collected for this study population as it is not routinely done. Graft versus Host Disease and treatment related toxicity is reported in the secondary outcome measure section.
Arm/Group | Intent-To-Treat
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study ended early as thymic shielding was found to be safe. Therefore, a new study was designed using thymic shielding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes